CLINICAL TRIAL: NCT00698100
Title: Vaccination of AJCC Stage IIB, IIC, III and IV Melanoma Patients With Human and Mouse Tyrosinase DNA Vaccines: A Phase I Trial to Assess Safety and Immune Response
Brief Title: Vaccination of AJCC Stage IIB, IIC, III and IV Melanoma Patients With Human and Mouse Tyrosinase DNA Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 99-122
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Melanoma; Skin
Keywords: DNA; HU & MOUSE; TYROSINASE
MeSH Terms: conditions — Melanoma

ARMS (2):
- 1 (Experimental): Patients will get human tyrosinase vaccination.
  Interventions: Biological: human tyrosinase
- 2 (Experimental): Patient will get mouse tyrosinase DNA vaccination.
  Interventions: Biological: mouse tyrosinase

INTERVENTIONS:
Biological: human tyrosinase — Patients will receive a total of 6 vaccinations. Each vaccination is given via the intramuscular route. Sites of injection should have intact lymphatic drainage. The vaccinations will be administered at three week intervals. Groups of six patients will be randomized at each dose level to receive either three immunizations with mouse tyrosinase followed by three immunizations with human tyrosinase or three immunizations with human tyrosinase followed by three immunizations with mouse tyrosinase
  Arms: 1
Biological: mouse tyrosinase — Patients will receive a total of 6 vaccinations. Each vaccination is given via the intramuscular route. Sites of injection should have intact lymphatic drainage. The vaccinations will be administered at three week intervals. Groups of six patients will be randomized at each dose level to receive either three immunizations with mouse tyrosinase followed by three immunizations with human tyrosinase or three immunizations with human tyrosinase followed by three immunizations with mouse tyrosinase
  Arms: 2

SUMMARY:
The overall goal of this study is to find out about the safety of injecting the genes (DNA) for human and mouse tyrosinase in patients with melanoma. There is no evidence yet that injection of tyrosinase DNA results in any clinical benefit. Tyrosinase is the substance found in melanoma cells that helps to produce their black color. The DNA used in this study was purified from bacteria which contains the gene for tyrosinase. DNA is material which contains the information needed to produce many substances in the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented malignant melanoma, American Joint Commission on Cancer (AJCC) stage IIB, IIC, III or IV. Patients free of disease after surgical resection will also be eligible.
* For all patients, pathology slides must be reviewed by the Memorial Hospital Department of Pathology for confirmation of melanoma diagnosis.
* Patients must be HLA-A0201 positive.
* Patients must be at least 18 years of age to be eligible and must be able to read the informed consent and give informed consent.
* Patients must have a Karnofsky performance status of at least 80.
* LDH < than or = to 2x upper limit of normal value; albumin > than or = to 3.5 mg/dl.
* A CBC prior to vaccination with WBC > or = to 3000, platelets > or = to 100,000.
* Patients must be free of detectable brain metastases.

Exclusion Criteria:

* Patients may not be receiving or have received chemotherapy, immunotherapy or radiation therapy within the previous 4 weeks. Patients must be fully recovered from any previous therapy or surgery.
* Patients may not have been previously immunized with vaccines containing tyrosinase or peptides derived from tyrosinase.
* Any medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to respond immunologically to vaccines is grounds for exclusion, at the discretion of the Principal Investigator or co-Principal Investigators.
* Patients who have preexisting retinal or choroidal eye disease will be excluded.
* Patients with serious underlying medical conditions, active infections requiring antimicrobial drugs, or active bleeding will be ineligible.
* Pregnant women or women who are less than 3 months post-partum are not eligible. Women who may yet bear children and sexually active men must be using appropriate contraception during the course of this study. Women of child-bearing potential must not be pregnant (negative BHCG within 2 weeks of vaccination) nor be nursing during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Is to determine the safety and immunogenicity of vaccination with the genes coding for mouse and human tyrosinase in patients. | conclusion of the study

SECONDARY OUTCOMES:
To evaluate antibody and CD8+ T cell responses to human tyrosinase after vaccination. | conclusion of the study
Is to observe the patients for evidence of any anti-tumor response, which is generated after vaccination. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jedd Wolchok, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org